CLINICAL TRIAL: NCT04904653
Title: Randomized Controlled and Single Blind Clinical Trial in Women With Breast Cancer and Axillary Lymphadenectomy, to Evaluate the Effectiveness of Hemopatch® in the Reduction of Post-surgical Serous Drainage
Brief Title: The Effectiveness of Hemopatch® in the Reduction of Post-surgical Serous Drainage
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Asociación De Cirujanos De Mama De Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HVST-HEMO-20
Record Dates: First submitted 2021-05-19; First posted 2021-05-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hemopatch; Breast Cancer; Axillary Lymphadenectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: After axillary node dissection, patients will be randomised to:
  * Hemopatch Group: Hemopatch (hemostatic device and surgical sealant) + suction drainage
  * Control group: no sealant (liquid, gel or patch) + suction drain
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemopatch Group: (Experimental): Hemopatch + suction drainage
  Interventions: Device: Hemopatch
- Control group (Other): No sealant (liquid, gel or patch) + suction drain
  Interventions: Other: Control group

INTERVENTIONS:
Device: Hemopatch — HEMOPATCH Sealing Hemostat ("HEMOPATCH") consists of a soft, thin, pliable, flexible pad of collagen derived from bovine dermis, coated with NHS-PEG (pentaerythritol polyethylene glycol ether tetra-succinimidyl glutarate).
  Due to its flexible structure, the application of HEMOPATCH to the site where hemostasis / sealing is desired is easily controlled. For differentiation, the non-coated side is marked with blue squares using a biocompatible colorant.
  HEMOPATCH is supplied in the following 3 sizes:
  * HEMOPATCH 27 x 27 mm
  * HEMOPATCH 45 x 45 mm
  * HEMOPATCH 45 x 90 mm
  Arms: Hemopatch Group:
Other: Control group — No sealant (liquid, gel or patch) + suction drain
  Arms: Control group

SUMMARY:
Hemopatch is an alternative to reduce morbidity associated with axillary lymphadenectomy surgery, possibly contributing to improved patient management, clinical outcomes, and hospital costs. We propose a multicenter, controlled, and randomized trial to study the efficacy of Hemopatch in reducing serous wound drainage.

ELIGIBILITY:
INCLUSION CRITERIA

Preoperative:

* Female gender
* Age ≥ 18 years
* Breast cancer N+
* Conservative Surgery: Lumpectomy or Quadrantectomy
* Berg levels 1-2 axillary lymphadenectomy

Intraoperative:

* Axillary incision separated from the incision for the breast lesion
* Placement of a closed low pressure suction drain in the axillary fossa
* Hemostasis and lymphostasis using clips, electrocautery, electric scalpel or bipolar coagulation

Postoperative:

- Patients with ≥ 10 axillary nodes removed

EXCLUSION CRITERIA

Preoperative:

* Mastectomy
* Previous radiation therapy
* Previous axillary emptying
* Liver pathology
* Diabetic decompensation: defined as any episode that has required medical attention in an emergency service or hospital admission; and also that which has required a modification of the patient's drugs, or an increase of more than 20% of the total daily dose.
* Known allergies to any component of Hemopatch (proteins of bovine origin or PEG)
* Psychiatric disorder that conditions the non-understanding of the questionnaire, or incapacitation of the patient to understand it
* Simultaneous participation in another clinical study
* PCR positive for SARS-CoV-2

Intraoperative:

* Level 3 axillary dissection (severe axillary involvement)
* Unexpected surgical contraindication
* Hemostasis and lymphostasis: ultrasonic techniques or other advanced energy techniques are excluded.
* Use of fibrin sealants (eg: Tisseel, Artiss, Tachosil), cyanoacrylate type adhesives (eg: Glubran-2) or other types of products (oxidized cellulose format, powders or gelatin sheets or collagen).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Total volume in milliliters (ml) of drainage | In the last 24 hours
  Total volume in milliliters (ml) of drainage: To be measured in the hospital every day before discharge, and collected daily after discharge with a follow-up of phone calls or patient diaries during hospital visits until extraction drain.

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery and Digestive System Service, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No